CLINICAL TRIAL: NCT04641572
Title: Application the Recommended Positions of the World Health Organization During Normal Childbirth and Its Effect on Maternal and Labor Outcomes
Brief Title: Different Positions During Childbirth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Howieda Fouly, Assistant professor, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Woman's health Hospital
Record Dates: First submitted 2020-07-05; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-10

CONDITIONS: Childbirth Process

STUDY DESIGN:
Intervention Model Description: Random selection based on the woman's preference for certain positions during her first stage of labor.
Who Masked: Participant, Care Provider
Masking Description: The researcher will use the simple randomize technique ( lottery withdrawal) to give the participants the right to pick up one of these positions through three letters will be written in three folded papers and put in an envelope, each letter will refer to a certain method. As soon as chosen of the letter the research will apply the chosen method and explain the benefits of that position/ technique for the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine position (No Intervention): group A ( control ) will follow the hospital routine positions either supine or lateral during labor
- Upright position (Experimental): Group B (intervention) will follow the Standing or walking, Squatting, Sitting, Hands /knees, and Kneeling, positions. Then the researcher will register the time ( minutes/hours) that will be taken and which will be more preferable by the participant.
  Interventions: Other: Choose comfortable position

INTERVENTIONS:
Other: Choose comfortable position — Standing or walking, Squatting, Sitting, Hands /knees, and Kneeling, positions will be taken by the participant during labor.Then the researcher will register the time ( minutes/hours) will be taken and which that will be more preferable by the participant
  Other Names: change position
  Arms: Upright position

SUMMARY:
To encourage the application the recommended positions of the World Health Organization during normal childbirth and its effect on maternal and labor outcomes

DETAILED DESCRIPTION:
To assess the effects of adopting upright positions (walking, sitting, standing) during first stage of labor.

To measure the effect of different individual positions on maternal-fetal outcomes.

To determine which position was more comfortable for women.

ELIGIBILITY:
Inclusion Criteria:

* aged > 18 years old with normal pregnancy, primiparas and multi-paras labor cases.

Exclusion Criteria:

* All high-risk associated factors (Hypertension- DM, Heart disease- renal disease) will be excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Childbirth process specific to females
Enrollment: 300 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
The maternal outcome. | Within labor process
  measure labor pain score in each position on pain scale
Newborn outcome | At 1 minute and 5 minutes after delivery.
  Measure the APGAR score of the newborn related to each position

SECONDARY OUTCOMES:
-Increase self-direction of participants through choosing the preferable position | Within labor process
  Register the most preferable positions during childbirth process
Improve women's satisfaction of childbirth experience | After childbirth process.
  measure woman's satisfaction after application of the upright position

CONTACTS AND LOCATIONS:
Overall Officials: Howieda Fouly, PhD, Principal Investigator — Woman's Health Hospital
Locations (1):
- Woman Health Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
The data only will be available for the study co-investigators.